CLINICAL TRIAL: NCT03822702
Title: An Alternative Perspective to Comprehend Handwriting Performance: Development and Applications of a Biomechanical Assessment and Biofeedback-training System for Handwriting (BABSH)
Brief Title: Biomechanical Assessment and Biofeedback-training System for Handwriting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A-ER-103-385
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Writing Learning Disability
Keywords: handwriting; kinetics; kinematics; handwriting difficulty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1st part:System development of Adult (No Intervention): No intervention. Subjects need to use 6 types of special pen to do the specific writing tasks for one hour.
  The same tasks will be ask to do again three days later.
- 1st part:System development of Child (No Intervention): No intervention. Subjects need to use 6 types of special pen to do the specific writing tasks for one hour.
  The same tasks will be ask to do again three days later.
- 2nd part:Handwriting Difficulty (No Intervention): No intervention. Subjects need to do the specific writing tasks and fine motor test for one hour with sensors on the hand. A handwriting screening questionnaire shall be filled.
- 3rd part: Biofeedback Training (Experimental): This program includes 1 hour pre-test, 8 times training and 1 hour post-test. For pre-test, subjects need to do the specific writing tasks and fine motor test for one hour. A handwriting screening questionnaire shall be filled.
  For post-test, the same procedure will be ask to do again about one and a half month later .
  After pre-test, eight times of Biofeedback Training will be asked. Each time will take 50 minutes, one or two times a week. All training will be completed in about one and a half month.
  Interventions: Other: Biofeedback Training
- 3rd part: Motor Training (Experimental): This program includes 1 hour pre-test, 8 times training and 1 hour post-test. For pre-test, subjects need to do the specific writing tasks and fine motor test for one hour. A handwriting screening questionnaire shall be filled.
  For post-test, the same procedure will be ask to do again about one and a half month later .
  After pre-test, eight times of Motor Training will be asked. Each time will take 50 minutes, one or two times a week. All training will be completed in about one and a half month.
  Interventions: Other: Motor Training
- 3rd part:Control Group (No Intervention): No intervention. Subjects need to do the specific writing tasks and fine motor test for one hour. A handwriting screening questionnaire shall be filled.
  The same procedure will be ask to do again about one and a half month later.

INTERVENTIONS:
Other: Biofeedback Training — Biofeedback training targeted to goals that are relevant to the handwriting skills for children by using a force acquisitional pen.
  Arms: 3rd part: Biofeedback Training
Other: Motor Training — Motor training targeted to goals that are relevant to the handwriting skills for children by using a personal designed motor training program.
  Arms: 3rd part: Motor Training

SUMMARY:
The purpose of this study is to investigate the real-time kinetics of handwriting regarding the design of the utensil and fine motor performances from biomechanical perspectives. It includes three parts.

The first part is an observational study design and the specific aim of the first part of the study is to establish a novel kinetic assessment system incorporated with Force Acquisition Pens (FAPs) designed with different barrel sizes and shapes for handwriting. The thorough calibration, examination of reliability and validity will be presented in this study.

The second part is also an observational study design and the specific aim of the second part of the study is to investigate the handwriting mechanisms using the kinetic assessment system incorporated with the motion capture system with children who have writing difficulties.

The third part is an interventional study design and the aim of this final part is to integrate the kinetic assessment system and the intervention concept to establish a Biomechanical Assessment and Biofeedback-training System for Handwriting (BABSH). Comparison of the intervention effect of the BABSH and traditional training for the children with handwriting difficulties will also be carried out in this part.

ELIGIBILITY:
Inclusion Criteria:

1. Able to use pen to write
2. Children volunteers must study in elementary schools

Exclusion Criteria:

- Handwriting problems are related to muscular, skeletal, nerve and brain damage or disease.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2016-05-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in the result of Chinese Handwriting Evaluation Form | baseline, 1.5 months
  A questionnaire about handwriting performance. Each item is rated on a five-point ordinal scale
Change in the total point score of three subtests of Bruininks-Oseretsky Test of Motor Proficiency, Second Edition (BOT-2) | baseline, 1.5 months
  These three subtests are 'fine motor precision (subtest-1) ', 'fine motor integration (subtest-2)' and 'manual dexterity (subtest-3)'.
  The raw scores of the three subtests were then transformed into point scores based on the BOT-2 manual. The total point scores of the three subtests will be analyzed. For subtest-1, the range of total point score is 0 to 41. For subtest-2, the range of total point score is 0 to 40. For subtest-3, the range of total point score is 0 to 45. Higher total point scores represent a better performance (outcome).
Change in the handwriting kinetic parameters | baseline, 1.5 months
  The kinetic parameters designed by measuring the real finger force applied on a force acquisitional pen.
Change in the handwriting kinematic parameters | baseline, 1.5 months
  The kinematic parameters designed by measuring the real hand motion using motion analysis system.

SECONDARY OUTCOMES:
Change in the pinch force | baseline, 1.5 months
  three types of pinch force were recorded by a pinch meter

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University, Tainan, Taiwan